CLINICAL TRIAL: NCT04735848
Title: Single Center Clinical Trial to Evaluate the Effect of Different Amounts of Iron Supplements on the Plasma Hepcidin Level in Non-anemic Iron-deficient Females
Brief Title: Plasma Hepcidin Response to Differently Dosed Iron Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pierre-Alexandre Krayenbuehl (Other)
Responsible Party: Sponsor-Investigator, Pierre-Alexandre Krayenbuehl, Research associate at the Clinic for Endocrinology, University of Zurich
Organization: University of Zurich (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Plasma hepcidin response
Record Dates: First submitted 2021-01-19; First posted 2021-02-03 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Iron Deficiency (Without Anemia)
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: The participants will take all three different doses of iron and will serve as there own control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 6mg iron-supplement (Experimental): All participants will be in this arm. Everyone will take all three different doses of iron-supplement (6mg; 30mg;60mg).
  Interventions: Dietary Supplement: Iron-supplement application
- 30mg iron-supplement (Experimental): All participants will be in this arm. Everyone will take all three different doses of iron-supplement (6mg; 30mg;60mg).
  Interventions: Dietary Supplement: Iron-supplement application
- 60mg iron-supplement (Experimental): All participants will be in this arm. Everyone will take all three different doses of iron-supplement (6mg; 30mg;60mg).
  Interventions: Dietary Supplement: Iron-supplement application
- Baseline (No Intervention): Baseline measurement

INTERVENTIONS:
Dietary Supplement: Iron-supplement application — The participants will take the corresponding amount of iron-supplement supervised at 8am.
  Arms: 30mg iron-supplement; 60mg iron-supplement; 6mg iron-supplement

SUMMARY:
The study participants will take 3 different doses of iron supplements at 8 am, on 3 different days. By taking blood samples in the morning and afternoon, the investigators will determine the effects of the iron supplements on plasma hepcidin and compare them to baseline plasma hepcidin values.

DETAILED DESCRIPTION:
15 healthy young women with non-anemic iron deficiency will participate in the study. On 4 different days the investigators will take two blood samples (one in the morning at 8 am, before the iron intake and one in the afternoon at 4 pm) to determine the plasma hepcidin level. The intake of the iron supplements will be at least 48 hours apart from each other, to exclude any impacts of the previous iron intake to the next measurement.

The participants will take the iron supplement supervised at 8 am after overnight fasting.

All blood samples will be performed for analysis of CRP and hepcidin. The investigators will measure the CRP in the blood sample to exclude any impacts of inflammation to the hepcidin measurement and use a CRP ≤5mg/l as a cut-off. If the CRP is higher than 5mg/l the investigators will exclude the measurement from our analyses and repeat the measurement at another day.

The first two blood samples will be taken at 8 am and at 4 pm on the same day and after overnight fasting to find the baseline hepcidin, the other blood samples will be taken at 8 am before the iron intake and at 4 pm also on the same day and also after overnight fasting.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Female gender
* Premenopausal
* Age > 18 years
* Regular menstrual cycle
* BMI in normal range (18-25kg/m2)
* Serum-ferritin ≤30ng/ml
* No anemia
* No intake of dietary supplements

Exclusion Criteria:

* Intake of dietary supplements
* Pregnancy
* Hypermenorrhea (> 80ml blood loss, or more than 5 unties/tampons per day)
* Anemia
* Serum-ferritin >30ng/ml
* BMI <18 kg/m2 or >25 kg/m2
* Chronic inflammatory disease
* Hypersensitivity to iron supplements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Plasma hepcidin change | The hepcidin measurement of all samples will be done after the last blood sample of the last participant is taken. Which is planed to be done up to 6 month from the first baseline visit.
  The investigators will measure the plasma hepcidin level of the patients in the morning at 8am, (right before the intake of the iron-supplement) as well as in the afternoon at 4pm. The investigators will also measure the plasma hepcidin level on a baseline day (at the same times), when the patients don't take any iron supplement. By these measurements the investigators will report the change in the plasma hepcidin level after the intake of an iron-supplement.

SECONDARY OUTCOMES:
Dose-response relationship between iron and hepcidin | The hepcidin measurement of all samples will be done after the last blood sample of the last participant is taken. Which is planed to be done up to 6 month from the first baseline visit.
  In addition, the investigators will estimate a linear relationship (slope) between the iron dose and the plasma hepcidin level, using dose as a continuous explanatory factor in the model. The investigators will report a dose dependent assessment of the plasma hepcidin level.

OTHER OUTCOMES:
Number of participants with side effects | The participants will be asked for side effects in the afternoon of the same day as the participants take the iron-supplement. The analysis of the reported side-effects is planed to be done up to 6 month from the first baseline visit.
  The investigators will analyze number the side effects named as nausea, abdominal pain or constipation, which occurred on the day of the iron-intake and were reported at the interview in the afternoon. The investigators will compare the amount of side-effects that occurred in each dosage group. The investigators expect a dose-dependent occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexandre Krayenbühl, Principal Investigator — University of Zurich
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland

REFERENCES:
- [Derived] Karczewski M, Simic S, Saleh L, Nowak A, Schubert MG, Moretti D, Swinkels DW, Beuschlein F, Suter PM, Krayenbuehl PA. The magnitude of the plasma hepcidin response to oral iron supplements depends on the iron dosage. Swiss Med Wkly. 2024 Feb 19;154:3635. doi: 10.57187/s.3635. PMID 38579297